CLINICAL TRIAL: NCT04949776
Title: New Strategies Based on Artificial Intelligence in Breast Cancer Screening Programs in Córdoba With Digital Mammography and Digital Breast Tomosynthesis. A Prospective Evaluation.
Brief Title: Artificial Intelligence in Breast Cancer Screening Programs
Acronym: AITIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AITIC
Record Dates: First submitted 2021-06-15; First posted 2021-07-02 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Screening
Keywords: breast cancer; artificial intelligence; Digital breast tomosynthesis; Mammography; Mass screening
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Double reading of all cases with and without Transpara software (Experimental): Double reading of all cases with and without Transpara software
  Interventions: Diagnostic Test: Mammograms

INTERVENTIONS:
Diagnostic Test: Mammograms — In the women participating in the study, two strategies for reading mammograms will be carried out:
  Strategy 1: Standard reading of the program. Double independent and non-consensual reading of all cases, without any artificial intelligence system (standard strategy).
  Strategy 2: Reading strategy based on the global Score granted by Transpara® (strategy based on artificial intelligence):
  * In studies with a Score <8 (studies with a low probability of cancer): They will not be evaluated by any radiologist.
  * In studies with a Score> 7 (studies with a high probability of cancer): double reading will be carried out, assisted by Transpara®.

SUMMARY:
The use of artificial intelligence software in breast screening (Transpara®) makes it possible to identify studies with a very low probability of cancer.

The hypothesis raised in this work is that reading strategies based on artificial intelligence (single or double reading only of cases with a score> 7 with Transpara®), allow reducing the workload of a screening program by more than 50 % with respect to the standard reading of the program (double reading of all cases without Transpara®), without presenting inferiority in terms of detection rates and recalls of the program, both with the use of 2D digital mammography and with the use of tomosynthesis or 3D mammogram.

ELIGIBILITY:
Inclusion criteria:

All women between 50 and 71 years of age (including women who reach that age in the year of appointment), in the Reina Sofía University Hospital district, invited to participate in the Breast Cancer Early Detection Program, that have been randomly assigned in the Hologic equipment (DM or DBT), and who agree to participate in the study by signing the informed consent form.

1. Women studied in the program during the established period and who have previously participated.
2. Women studied in the program for the first time in the established period.

Exclusion Criteria:

1. Women invited to the program who do not agree to participate in the research study by signing the informed consent form.
2. Women with breast prostheses.
3. Women with signs or symptoms of suspected breast cancer.

Ages: 50 Years to 71 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women participating in the regular Breast Cancer Early Detection Program in Cordoba
Enrollment: 31301 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Assessment of Workload of each strategy | In the middle of the study, at 1 year.
  The workload of each strategy shall be assessed by multiplying the average time for a reading of that strategy by the total number of readings of that strategy.
  The average reading time of a case in each strategy shall be calculated from the measurement of the individual reading time in a sample of 500 cases in each strategy.
Assessment of Workload of each strategy | At the end of the study, at 2 years.
  The workload of each strategy shall be assessed by multiplying the average time for a reading of that strategy by the total number of readings of that strategy.
  The average reading time of a case in each strategy shall be calculated from the measurement of the individual reading time in a sample of 500 cases in each strategy.
Detection rate | In the middle of the study, at 1 year.
  Proportion of women diagnosed with breast cancer among those screened.
Detection rate | At the end of the study, at 2 years.
  Proportion of women diagnosed with breast cancer among those screened.
Recall or referral rate | In the middle of the study, at 1 year.
  Proportion of women who, after the screening test, are referred to the breast diagnosis unit.
Recall or referral rate | At the end of the study, at 2 years.
  Proportion of women who, after the screening test, are referred to the breast diagnosis unit.

SECONDARY OUTCOMES:
Positive predictive value of referrals | In the middle of the study, at 1 year.
  Proportion of women diagnosed with breast cancer among those referred to the hospital.
Positive predictive value of referrals | At the end of the study, at 2 years.
  Proportion of women diagnosed with breast cancer among those referred to the hospital.
Positive predictive value of biopsies | In the middle of the study, at 1 year.
  Proportion of women with breast cancer among all women undergoing biopsy.
Positive predictive value of biopsies | At the end of the study, at 2 years.
  Proportion of women with breast cancer among all women undergoing biopsy.
Positive predictive value of Transpara® scores | In the middle of the study, at 1 year.
  Proportion of breast cancers diagnosed among women with a given score.
Positive predictive value of Transpara® scores | At the end of the study, at 2 years.
  Proportion of breast cancers diagnosed among women with a given score.

CONTACTS AND LOCATIONS:
Overall Officials: Esperanza Elias Cabot, MD, Principal Investigator — Hospital Universitario Reina Sofia de Cordoba
Locations (1):
- Hospital Universitario Reina Sofia, Córdoba, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
The database and the protocol Will be shared after the trial is published.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the trial is published.
Access Criteria: Upon request to the principal investigator.

REFERENCES:
- [Background] Raya-Povedano JL, Romero-Martin S, Elias-Cabot E, Gubern-Merida A, Rodriguez-Ruiz A, Alvarez-Benito M. AI-based Strategies to Reduce Workload in Breast Cancer Screening with Mammography and Tomosynthesis: A Retrospective Evaluation. Radiology. 2021 Jul;300(1):57-65. doi: 10.1148/radiol.2021203555. Epub 2021 May 4. PMID 33944627
- [Background] Rodriguez-Ruiz A, Lang K, Gubern-Merida A, Broeders M, Gennaro G, Clauser P, Helbich TH, Chevalier M, Tan T, Mertelmeier T, Wallis MG, Andersson I, Zackrisson S, Mann RM, Sechopoulos I. Stand-Alone Artificial Intelligence for Breast Cancer Detection in Mammography: Comparison With 101 Radiologists. J Natl Cancer Inst. 2019 Sep 1;111(9):916-922. doi: 10.1093/jnci/djy222. PMID 30834436
- [Background] Rodriguez-Ruiz A, Lang K, Gubern-Merida A, Teuwen J, Broeders M, Gennaro G, Clauser P, Helbich TH, Chevalier M, Mertelmeier T, Wallis MG, Andersson I, Zackrisson S, Sechopoulos I, Mann RM. Can we reduce the workload of mammographic screening by automatic identification of normal exams with artificial intelligence? A feasibility study. Eur Radiol. 2019 Sep;29(9):4825-4832. doi: 10.1007/s00330-019-06186-9. Epub 2019 Apr 16. PMID 30993432
- [Background] Rodriguez-Ruiz A, Krupinski E, Mordang JJ, Schilling K, Heywang-Kobrunner SH, Sechopoulos I, Mann RM. Detection of Breast Cancer with Mammography: Effect of an Artificial Intelligence Support System. Radiology. 2019 Feb;290(2):305-314. doi: 10.1148/radiol.2018181371. Epub 2018 Nov 20. PMID 30457482
- [Background] Yala A, Schuster T, Miles R, Barzilay R, Lehman C. A Deep Learning Model to Triage Screening Mammograms: A Simulation Study. Radiology. 2019 Oct;293(1):38-46. doi: 10.1148/radiol.2019182908. Epub 2019 Aug 6. PMID 31385754
- [Background] Sasaki M, Tozaki M, Rodriguez-Ruiz A, Yotsumoto D, Ichiki Y, Terawaki A, Oosako S, Sagara Y, Sagara Y. Artificial intelligence for breast cancer detection in mammography: experience of use of the ScreenPoint Medical Transpara system in 310 Japanese women. Breast Cancer. 2020 Jul;27(4):642-651. doi: 10.1007/s12282-020-01061-8. Epub 2020 Feb 12. PMID 32052311
- [Background] Le EPV, Wang Y, Huang Y, Hickman S, Gilbert FJ. Artificial intelligence in breast imaging. Clin Radiol. 2019 May;74(5):357-366. doi: 10.1016/j.crad.2019.02.006. Epub 2019 Mar 18. PMID 30898381